CLINICAL TRIAL: NCT02093611
Title: Study to Examine the Effects of ATP Supplementation on Muscle Excitability and Reaction Time During and Following a Repeated Sprint Bout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: University of Tampa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MTI2013-CS04
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Muscle Fatigue Caused by Repetitive Muscle Exercise
MeSH Terms: interventions — Adenosine Triphosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): This arm will serve as the placebo supplementation.
  Interventions: Dietary Supplement: Placebo
- ATP (Active Comparator): This arm will serve as the treatment intervention, ATP
  Interventions: Dietary Supplement: ATP

INTERVENTIONS:
Dietary Supplement: Placebo
  Other Names: Placebo Comparator
  Arms: Placebo
Dietary Supplement: ATP — 400 mg of ATP
  Other Names: Peak ATP
  Arms: ATP

SUMMARY:
We hypothesize that adenosine-5'-triphosphate (ATP) supplementation will be able to enhance motor unit recruitment while simultaneously blunting the decline in power and reaction time that is typically seen during repetitive sprints. This will give researchers a better understanding of the mechanism by which ATP supplementation can augment power, especially under high fatiguing conditions.

DETAILED DESCRIPTION:
Healthy participants of similar training status as previously tested will be enrolled into the study. The participants will be randomly assigned to either placebo supplementation or to 400 mg ATP per day for 14 days. The supplements will be taken in the morning and the last dose will be taken 30 min prior to testing on the last day. Testing will be performed at baseline and after the 14 days of supplementation. Ten successive sprints will be conducted on the Wingate apparatus as this has been previously demonstrated to decrease muscle excitability. After the sprints, muscle excitability, reaction time, and vertical jump power will be measured. In addition a blood sample will be obtained before and after supplementation and complete blood hematology and chemistry analyses will be performed. It is expected that ATP supplementation may help maintain muscle excitability and power after the successive sprint sessions.

ELIGIBILITY:
Inclusion Criteria:

* Agree to eating a diet approved by a registered dietician consisting of the following by caloric percentages: 15-20% protein, 44-55% carbohydrate, and 25-30% fat.
* Must not have taken performance enhancing supplements for at least 3 months prior to the study start,
* Must be a non-smoker.
* Must not be taking amino acid supplements.
* Must not be using anabolic or catabolic hormones.
* Must not be taking any medications known to influence variables to be measured in the study.

Exclusion Criteria:

* Will not agree to eating a diet approved by a registered dietician consisting of the following by caloric percentages: 15-20% protein, 44-55% carbohydrate, and 25-30% fat.
* Has taken performance enhancing supplements for at least 3 months prior to the study start,
* Is currently a non-smoker.
* Is currently taking amino acid supplements.
* Is currently using anabolic or catabolic hormones.
* Is currently taking medications known to influence variables to be measured in the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Muscle Excitability | Day 14
  Muscle excitability will be measured using Delsys Wireless Electromyography (EMG) sensors.

SECONDARY OUTCOMES:
Power | Day 14
  Muscle power will be measured using the Wingate and vertical jump power measures.

OTHER OUTCOMES:
Reaction Time | Day 14
  Reaction time will be measured using a Dynavision apparatus.
Blood Biochemical Analyses | Day 14
  Blood chemistries and hematology will be measured after the 14 days of supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Study Director — Metabolic Technologies Inc.
Locations (1):
- Jacob M Wilson, PhD, Tampa, Florida, United States